CLINICAL TRIAL: NCT05443581
Title: The Effect of Vegetarian Diet on Patients With Metabolic Associated Fatty Liver Disease：A Randomized Clinical Trial
Brief Title: The Effect of Vegetarian Diet on Patients With Metabolic Associated Fatty Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XH-22-004
Record Dates: First submitted 2022-05-23; First posted 2022-07-05 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2023-11

CONDITIONS: Metabolism and Nutrition Disorder; Liver Diseases; Obesity; Diet, Healthy
Keywords: Metabolism associated fatty liver disease; Obesity; Vegetarian diet; diet intervention
MeSH Terms: conditions — Nutrition Disorders; Liver Diseases; Obesity | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participations in this group are required to follow a healthy vegetarian diet （avoid meat, poultry, fish, dairy） during the 24-weeks trail.
  Daily energy intake = BMR(basal metabolic rate) × 1.25-500kcal；BMR = 370 + 21.6 × Lean body mass(kg) Requirements of energy supply ratio: protein 15%-20%; fat 20%-25%; carbohydrate 50%-60%.
  Interventions: Behavioral: dietary intervention
- Control group (Active Comparator): Participations in this group are required to follow a healthy omnivorous diet (No restriction on food sources) during the 24-weeks trail.
  Daily energy intake = BMR × 1.25-500kcal；BMR = 370 + 21.6 × Lean body mass(kg) Requirements of energy supply ratio: protein 15%-20%; fat 20%-25%; carbohydrate 50%-60%.
  Interventions: Behavioral: dietary intervention

INTERVENTIONS:
Behavioral: dietary intervention — Dietary guidance will be given to participants through monthly face-to-face interviews and biweekly telephone calls to change their dietary structure and energy intake.

SUMMARY:
In this study, 18-60 years old patients with metabolic associated fatty liver disease（MAFLD） will be recruited to test the intervention effect of vegetarian diet. This randomized clinical trial randomized individuals to a healthy vegetarian diet or a healthy omnivorous diet for 24 weeks. At the baseline and after the 24week intervention, the clinical manifestations of MAFLD, obesity levels, indices for glucose and lipid metabolism parameters, results of questionnaire and fecal samples will be collected and analyzed.

DETAILED DESCRIPTION:
Dietary control remains an important way for nutritional intervention of metabolic related fatty liver disease. However, studies shows that patients have low compliance to the traditional diet. The topic proposed based on previous studies，recruiting of 220 obesity patients with metabolic associated fatty liver disease aged 18-60. After the informed consent, they will be randomly divided into intervention group and control group, intervention group will be given healthy vegetarian diet intervention and the control group given healthy omnivorous diet. Both diets are in line with the principles of fatty liver treatment. Interventions consisted primarily of face-to -face interview monthly and online interview every 2 weeks, which will be performed by professional dietitians. All participants were asked not to alter their exercise patterns during the study period. The primary outcome was the weight of fat mass after 24 weeks intervention. Secondary outcomes included imaging findings (B-ultrasonic examination and Fibroscan) of MAFLD, liver function, anthropometric measures, plasma lipid and glucose levels. At the meantime, serum oxidative stress indices, results of compliance survey and metabolites of Intestinal flora will be collected and analyzed. Through the above detection of the indicators related to MAFLD and obesity, it is explored whether the vegetarian diet can be an efficient and feasible way to the nutritional therapy of MAFLD.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed as fatty liver, and BMI≥24.0kg/m²;
2. 18-60 years old;
3. Have not received drug treatment if having hyperglycemia, hyperlipidemia and high uric acid ;
4. No antibiotics in the last 1 month;
5. The guardian's informed consent;

Exclusion Criteria:

1. Have received drug treatment of fatty liver disease within three months;
2. Patients with with liver cirrhosis, viral hepatitis and other liver diseases;
3. Patients with serious heart, lung, kidney diseases and patients with cancer;
4. Pregnant and nursing women;
5. Other conditions that may affect the results of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
The primary outcome was the weight of fat mass after 24 weeks intervention. | 24 weeks
  Weight loss, especially the reduction of body fat mass, is the most important treatment for the prevention and treatment of MAFLD and its complicationsIn our study, we will measure weight of fat mass using a body composition analyzer (Biospace Inbody 720, Korea) at the baseline and after 24-week intervention. The difference in the weight of fat mass after intervention between the two groups is the primary outcome.

SECONDARY OUTCOMES:
Results of B-ultrasonic examination and Fibroscan examination | 24 weeks
  Imaging examination results are an important basis for the clinical diagnosis of NAFLD, which can show the degree of hepatic steatosis and hepatic fibrosis. Imaging findings of MAFLD will be measured and compared at the baseline and end of our study.
The changes of serum alanine aminotransferase (ALT) at week 24 intervention from the baseline | 24 weeks
  Hepatic steatosis is often accompanied by changes in hepatic enzymes.
The changes of serum aspartate aminotransferase (AST) at week 24 intervention from the baseline | 24 weeks
  Hepatic steatosis is often accompanied by changes in hepatic enzymes.
24-week weight change | 24 weeks
  The 24-week intervention is expected to bring weight loss. We will compare the weight loss between the two groups

OTHER OUTCOMES:
The Results of compliance survey will be collected every month. | 24 weeks
  We have designed a compliance scale to evaluate the compliance , which may be important to advise the nutritionists and doctors about the prevention and treatment of MAFLD.
The difference of serum superoxide dismutase (SOD) level between two groups after 24-week intervention | 24 weeks
  Cause vegetarian diet may contain more phytochemicals and less saturated fat and cholesterol due to the plant-based nature of the diet, resulting in better metabolic status and milder metabolic burden,we have presumed that the serum SOD level be different between two groups at the end of study.
The difference of metabolites of Intestinal flora between two groups after 24-week intervention. | 24 weeks
  The fecal samples before and after the intervention to examine the effect of vegetarian diets on gut microbiota metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Xiuhua Shen, Professor, Study Chair — Xinhua Hospital Afflicated to Shanghai Jiaotong University of Medicin
Locations (1):
- Department of Clinical Nutrition, Xinhua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No